CLINICAL TRIAL: NCT04650646
Title: Cardiovascular Effects of Exercise-related Hypoglycaemia in Patients With Type 1 Diabetes
Brief Title: Cardiovascular Effects of Exercise-related Hypoglycaemia in Patients With Type 1 Diabetes (Hypo Heart Exercise)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Tina Vilsbøll, Professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-20023688
Record Dates: First submitted 2020-11-12; First posted 2020-12-02 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 1; Arrhythmia
Keywords: Type 1 diabetes; Cardiovascular disease; Hypoglycaemia; Exercise-related hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Arrhythmias, Cardiac; Cardiovascular Diseases; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoglycaemic clamp i combination with exercise (Experimental): A 180 minutes hyperinsulinaemic euglycaemic-hypoglycaemic clamp in combination with an exercise session. The participants will be monitored with Holter-ECG throughout the entire clamp and plasma glucose will be measured every 5 minutes. Blood samples will be drawn and analysed for changes in electrolytes, counterregulatory hormones, coagulation status, inflammation, endothelial damage and oxidative stress.
  Interventions: Other: Exercise-related hypoglycaemia
- Hypoglycaemic clamp in combination with bed rest (Experimental): A 180 minutes hyperinsulinaemic euglycaemic-hypoglycaemic clamp in combination with bed rest. The participants will be monitored with Holter-ECG throughout the entire clamp and plasma glucose will be measured every 5 minutes. Blood samples will be drawn and analysed for changes in electrolytes, counterregulatory hormones, coagulation status, inflammation, endothelial damage and oxidative stress.
  Interventions: Other: Hypoglycaemia under resting conditions

INTERVENTIONS:
Other: Exercise-related hypoglycaemia — Hypoglycaemia induced by intravenous insulin and exercise on a vertical cycle ergometer.
  Arms: Hypoglycaemic clamp i combination with exercise
Other: Hypoglycaemia under resting conditions — Hypoglycaemia induced by intravenous insulin during bed rest.
  Arms: Hypoglycaemic clamp in combination with bed rest

SUMMARY:
Patients with type 1 diabetes are recommended to perform at least 150 minutes of accumulated physical activity each week, however fear of hypoglycaemia is a well-known barrier to exercise in these patients. Previous experimental studies have almost exclusively focused on investigating cardiovascular effects of hypoglycaemia under resting conditions, however other underlying circumstances prior to or during a hypoglycaemic event, (e.g. exercise) are rarely discussed in the literature but might, nevertheless, be of significant clinical importance.

In this study, the investigators aim to investigate the QT interval dynamics and prothrombotic factors during exercise-related hypoglycaemia in comparison with hypoglycaemia under resting conditions, in patients with type 1 diabetes.

Fifteen patients with type 1 diabetes will be recruited for a crossover study including two test days, a combined euglycaemic- hypoglycaemic clamp combined with an exercise session and an euglycaemic- hypoglycaemic clamp during bed rest, respectively. Furthermore, the participants will be schedueled for a 24-hours followup visit after each test day for the purpose of investigating prolonged prothrombotic effects of hypoglycaemia. Patients will be randomised 1:1 to start with the combined exercise-clamp or the resting-clamp. The two test days will be separated by at least 4 weeks to minimise carry-over effects. A group of fifteen healthy individuals with normal glucose tolerance matched for age, gender and body mass index, will be recruited for a single blood test aiming to compare baseline coagulation status with patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Type 1 diabetes diagnosed according to the criteria of the World Health Organization (WHO)
* Age ≥ 18 years
* Insulin treatment for ≥1 year

Exclusion Criteria:

* Arrhythmia diagnosed prior to the screening visit.
* Ischaemic heart disease or myocardial infarction diagnosed prior to the screening visit.
* Implantable cardioverter defibrillator (ICD) or pacemaker at the time of inclusion
* Heart failure (left ventricular ejection fraction <45%) diagnosed prior to the screening visit.
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* ECG with left or right bundle branch block diagnosed prior to the screening visit.
* Thyroid dysfunction (except for well-regulated levothyroxine-substituted myxoedema)
* Anaemia (male: haemoglobin <8.0; female: haemoglobin <7.0 mmol/l)
* Treatment with anticoagulant or antiplatelet treatment.
* Bleeding disorder diagnosed prior to the screening visit.

Withdrawal criteria

- The participants may withdraw at will at any time

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Hypoglycaemia and QTc interval prolongation | 0-180minutes
  Mean QTc interval prolongation from baseline during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.

SECONDARY OUTCOMES:
Key secondary outcome: Hypoglycaemia and coagulation and fibrinolysis | 0-24hours
  Differences in whole blood coagulability and fibrinolysis (measured by thrombelastography) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and QT dispersion (QTd) | 0-180minutes
  Differences in QTd, during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions
Hypoglycaemia and heart rate variability (HRV) | 0-180minutes
  Changes in sympathetic/parasympathetic balance (measured by HRV) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and bradycardia | 0-180minutes
  Differences in non-clinically significant bradycardia (≤45 bpm for 5 seconds) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and ectopic beats | 0-180minutes
  Differences in number of atrial ectopic beats (prematurity threshold 30%) and ventricular premature beats respectively, during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and endothelial activation and damage | 0-24hours
  Differences in plasma markers of endothelial activation and damage (ng/ml) (including Syndecan-1, Soluble thrombomodulin and PECAM-1) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and vascular oxidative stress | 0-24hours
  Differences in markers of vascular oxidative stress (tetrahydrobiopterin/dihydrobiopterin ratio, dehydroascorbic acid/ascorbic acid ratio, asymmetric dimethylarginine/arginine ratio, malondialdehyde) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and electrolytes | 0-180minutes
  Differences in electrolyte concentrations including potassium and ionised calcium during exercise-related hypoglycaemia compared insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and counterregulatory hormonal response | 0-180minutes
  Differences in hormonal response (plasma glucagon, cortisol, catecholamines and growth hormone) during exercise-related hypoglycaemia compared insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and markers of inflammation | 0-24hours
  Differences in inflammatory response (including interleukin 6 and TNFα) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and inflammation | 0-24hours
  Differences in High-sensitive C-reactive peptide (HsCRP) during exercise-related hypoglycaemia compared to insulin-induced hypoglycaemia under resting conditions.
Hypoglycaemia and continuous glucose monitoring (CGM) accuracy | 0-180min
  Differences in mean absolute relative difference (MARD) between Dexcom G6®, Abbot Flash Libre® and Yellow Springs Instrument (YSI) reference throughout both experimental days.
Type 1 diabetes, healthy controls and coagulability | 0minutes
  Differences in whole blood coagulability and fibrinolysis (measured by thrombelastography) between patients with type 1 diabetes and healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD, DMSc, Principal Investigator — Steno diabetic centre (SDCC)
Locations (1):
- Clinical Research, Steno Diabetes Center Copenhagen-Gentofte, Copenhagen, Denmark